CLINICAL TRIAL: NCT05894824
Title: An Open Label, Single-arm, Multicenter Phase Ib/II Study to Evaluate the Safety and Efficacy of T-Dxd in Combination With Ramucirumab as a 2nd Line in Patients With HER2 Low Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma
Brief Title: T-Dxd in Combination With Ramucirumab as HER2 Low Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Sun Young Rha, MD, Ph.D, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-0392
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer; Gastroesophageal Junction (GEJ) Cancer
Keywords: HER2 gastric cancer, T-Dxd, Ramucirumab
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms | interventions — Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm, Trastruzumab deruxtecan, Ramucirumab (Other): Single arm, Trastruzumab deruxtecan, Ramucirumab
  Interventions: Drug: T-Dxd(Trastuzmab deruxtecan), Ramucirumab

INTERVENTIONS:
Drug: T-Dxd(Trastuzmab deruxtecan), Ramucirumab — Phase Ib will use a standard 3+3 scheme with the planned doses of T-DXd (4.4~6.4 mg/kg) once every 3 weeks in combination with Ramucirumab 8mg/kg administered once every 2 weeks.
  * Dosing Regimen
    * Trastruzumab deruxtecan : One IV infusion every 3 weeks on Day 1 of each 21-day cycle
    * Ramucirumab : One IV infusion on every 2 weeks on Day 1,15 of each 28-day cycle
  Other Names: Enhertu, Cyramza

SUMMARY:
This is a Phase Ib/II study to identify the RP2D of T-DXd combination with Ram and to assess the safety and clinical efficacy of this combined treatment in advanced gastric cancer. The study will be conducted in two parts: Phase Ib dose escalation study to determine the MTD and RP2D of T-DXd combination and Ram, and Phase II to further evaluate the safety and tolerability of T-DXd combinations with Ram at the RP2D and determine anti-tumor activity.

DETAILED DESCRIPTION:
This is a Phase Ib/II study to identify the RP2D of T-DXd combination with Ram and to assess the safety and clinical efficacy of this combined treatment in advanced gastric cancer after first-line treatment. The study will be conducted in two parts: Phase Ib dose escalation study to determine the MTD and RP2D of T-DXd combination and Ram, and Phase II to further evaluate the safety and tolerability of T-DXd combinations with Ram at the RP2D and determine anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent and has signed the appropriate weitten informed consent form(ICF) prior to performance of any trial activityes.
2. Eligible male and female subjects aged ≥19 years.
3. Histologically or cytologically proven metastatic or locally advanced HER2 low gastric or GEJ adenocarcinoma: The definition of HER2 low is 1+ by immunohistochemistry (IHC) or 2+ by IHC and without HER2 gene amplification (negative by in situ hybridization[ISH]).
4. Progressed after 1st line palliative treatment. Adjuvant chemotherapy will be counted as 1st line treatment if the cancer has recurred within 6 months of completion of adjuvant chemotherapy.
5. Has measurable or evaluable disease as determined by RECIST ver 1.1.
6. ECOG performance status of 0 -1 at trial entry.
7. Life expectancy ≥12 weeks as judged by the Investigator.
8. Has LVEF ≥ 50% by either echocardiogram (ECHO) or multigated acquisition (MUGA) scan within 28 days before enrollment.
9. Adequate baseline organ function defined as:

   * Absolute neutrophil count ≥1500/mm3
   * Platelets ≥100,000/mm3
   * Hemoglobin ≥9.0 g/dL
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0 × upper limit of normal (ULN) of the study site (or ≤5.0 × ULN in patients with liver metastases)
   * Total bilirubin ≤1.5 × ULN - Serum albumin ≥2.5 g/dL
   * Creatinine ≤1.5 × ULN or creatinine clearance (either measured value or estimated value using the Cockcroft-Gault equation) >40ml/min - Urinary protein ≤1+ on dipsick or routine urinalysis - INR and PTT/aPTT ≤1.5 × ULN 10. Adequate treatment washout period before randomization/enrollment. - Major Surgery ≥ 4 weeks - Radiation Therapy including palliative stereotactic radiation therapy to chest ≥ 4 weeks
   * Anti-Cancer chemotherapy [Immunotherapy (non-antibody based therapy)] ≥ 3 weeks

11. Evidence of post-menopausal status or negative serum pregnancy test for females of childbearing potential who are sexually active with a non-sterilized male partner.

12. Female patients of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception from the time of screening and must agree to continue using such precautions for 7 months after the last dose of IMP.

13. Non-sterilized male patients who are sexually active with a female partner of childbearing potential must use a condom with spermicide from screening to 4 months after the final dose of IMP. 14. Female subjects must not donate, or retrieve for their own use, ova from the time of enrollment and throughout the study treatment period, and for at least 7 months after the final study drug administration

Exclusion Criteria:

1. Anticancer treatment within 14 days before the start of trial treatment.
2. Major surgery within 28 days before the start of trial treatment.
3. Have received more than 2 prior lines of chemotherapy.
4. Grade ≥ 2 peripheral neuropathy.
5. Multiple primary malignancies within 3 years.
6. Participants with a medical history of myocardial infarction within 6 months before treatment, symptomatic CHF (New York Heart Association Class II to IV), unstable angina pectoris, clinically important cardiac arrhythmias, or a recent (< 6 months) cardiovascular event, including myocardial infarction, unstable angina pectoris, and stroke.
7. Corrected QT interval (QTcF) prolongation to > 470 msec (females) or >450 msec (males) based on an average of the screening triplicate 12-lead ECG.
8. Gastrointestinal perforation or fistula or any Grade 3-4 bleeding within 3 months of first dose of protocol therapy; or any arterial thromboembolic event, significant gastro-intestinal bleeding or any significant venous thromboembolism within 3 months before treatment
9. History of (non-infectious) ILD / pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
10. Lung criteria: A. Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder. B. Any autoimmune, connective tissue or inflammatory disorders C. Prior pneumonectomy
11. Has known active CNS metastases and/or carcinomatous meningitis.
12. Has substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions that may, in the opinion of the investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
13. Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms.
14. Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals.
15. Active primary immunodeficiency, known uncontrolled active HIV infection or active hepatitis B or C infection, such as those with serologic evidence of viral infection within 28 days of Cycle 1 Day 1. 16. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. 17. Receipt of live, attenuated vaccine (mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first dose of trastuzumab deruxtecan. Note: Patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of IMP. 18. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤ 1 or baseline. 19. Known allergy or hypersensitivity to study treatment or any of the study drug excipients.

20. History of severe hypersensitivity reactions to other monoclonal antibodies.

21. Pregnant or breastfeeding female patients, or patients who are planning to become pregnant.

22. Otherwise inappropriate for this study in the investigator's or sub-investigator's opinion.

23. Cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis.

24. Serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to first dose of protocol therapy.

25. The patient is receiving chronic antiplatelet therapy, including dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted.

26. The patient has uncontrolled or poorly-controlled hypertension (>160 mmHg systolic or > 100 mmHg diastolic for >4 weeks) despite standard medical management.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
RP2D | within first 6 weeks of treatment
  Maximum Tolerated dose (MTD) and Recommended phase 2 dose as determined by Dose limiting Toxicity (DLT).
PFS rate at 24 weeks | within first 2 4weeks of treatment
  Defined as the time from start of study treatment until the date of objective disease progression or death (by any cause in the absence of disease progression) Progression is defined in accordance with the RECIST v1.1 criteria. Determination of PFS rate at 24 weeks.

SECONDARY OUTCOMES:
Overall Survival (OS) | 6 months after the last treatment of the last subject
  Defined from the date of treatment assignment until the date of death due to any cause. Any participant not known to have died at the time of analysis will be censored based on the last recorded date on which the participant was known to be alive.
Objective Response Rate (ORR) | 6 months after the last treatment of the last subject
  Defined as the proportion of participants with measurable disease who achieve complete response(CR) or partial response(PR), as determined by the Investigator per RECIST v1.1. Data obtained up until disease progression, or the last evaluable assessment in the absence of progression, will be included in the assessment of ORR. Confirmatory scan is needed for the patients with CR or PR after 4 weeks of the first response. Participants who discontinue treatment without progression, receive a subsequent therapy, and then respond, will not be included as responders in the ORR.
Disease Control Rate (DCR) | 6 months after the last treatment of the last subject
  Defined as the percentage of participants who have a confirmed CR or PR or who have SD (without subsequent cancer therapy) after the date of treatment assignment.
Duration of Response (DoR) | 6 months after the last treatment of the last subject
  Defined as the percentage of participants who have a confirmed CR or PR or who have SD (without subsequent cancer therapy) after the date of treatment assignment.
Progression-free survival (PFS) | 6 months after the last treatment of the last subject
  Defined as time from the date of treatment assignment until progression per RECIST v1.1 as assessed by the Investigator, or death due to any cause. Participants who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment from their last evaluable RECIST v1.1 assessment.
adverse events categorized in accordance with CTCAE 5.0 Criteria. | 6 months after the last treatment of the last subject
  Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: SUN YOUNG RHA, Principal Investigator — Yonsei Cancer Center, Yonsei University College of Medicine
Locations (1):
- Sun Young Rha, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No